CLINICAL TRIAL: NCT06392893
Title: Evaluation of the Beneficial Health Effects of an Additive-free Meat Product in Healthy Subjects (HIPOCARNE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Hipocarne UMU 550/2023
Record Dates: First submitted 2024-04-16; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Inflammation; Oxidative Stress; Food Toxicity
Keywords: Additives; Allergens; Cooked ham; Cooked turkey breast; Inflammation; Oxidation; Nitrates; Gut microbiota
MeSH Terms: conditions — Inflammation | interventions — Meat Products; Allergens

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, controlled, unicentric trial with two parallel arms depending on the product consumed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Consumption of an additive and allergen-free cooked ham or cooked turkey breast.
  Quantity: 100 grams.
  Consumption time: 6 days a week during 5 weeks.
  Interventions: Combination Product: Meat product without additives and allergens
- Control (Placebo Comparator): Consumption of a commercial cooked ham or cooked turkey breast.
  Quantity: 100 grams.
  Consumption time: 6 days a week during 5 weeks.
  Interventions: Combination Product: Commercial meat product

INTERVENTIONS:
Combination Product: Meat product without additives and allergens — Baseline time: Measurement of anthropometric parameters and inflammatory and oxidative markers in blood, faeces and urine.
  Consumption of meat products without additives and allergens (6 days a week; 5 weeks).
  Final time: Measurement of anthropometric parameters and inflammatory and oxidative markers in blood, faeces and urine.
  Arms: Intervention
Combination Product: Commercial meat product — Baseline time: Measurement of anthropometric parameters and inflammatory and oxidative markers in blood, faeces and urine.
  Consumption of commercial meat products (6 days a week; 5 weeks).
  Final time: Measurement of anthropometric parameters and inflammatory and oxidative markers in blood, faeces and urine.
  Arms: Control

SUMMARY:
The purpose of this research is to test the hypothesis that the consumption of meat products without additives, in comparison with their analogues with additives, could be beneficial in terms of modifying health markers. A 5-week clinical trial with two parallel arms will be performed with two parallel arms. Changes in different serum biomarkers of lipid metabolism, glucose, oxidative stress and inflammation will be analysed. Biomarkers related to digestive health, such as short chain fatty acid (SCFA) production and impact on the gut microbiota, will also be evaluated. Finally, factors such as body mass index (BMI), body fat percentage and markers of exposure to additives will be measured.

DETAILED DESCRIPTION:
One of the most discussed reasons for reducing meat consumption is its additive content. Additives are compounds added to food products to preserve their technological properties, to avoid contamination by microorganisms, regulate acidity, and even act as thickeners, emulsifiers, and stabilisers. However, there is some controversy over the actual health effects of additives in meat products, as their long-term effect has not been studied for many of them. On the other hand, not all additives have the same effect, as for antioxidants such as sodium citrate (E-331) and sodium erythorbate (E-316), as well as acidity regulators such and triphosphates (E-451) no side effects or significant toxicity have been reported on healthy individuals. However, other additives such as carrageenans (E-407) have been associated with intestinal inflammation and inflammatory bowel diseases by several animal studies. Negative effects have also been found for sodium nitrite (E-250), which can lead to the formation of carcinogenic N-nitrosamines.

Due to the rising concern about additives in meat products, it is of particular interest to identify the possible health effects of a processed meat product without additives and allergens. Therefore, the hypothesis of this study is that the production of additive-free meat products may be of interest to the consumers and may have a beneficial effect on their health.

To confirm this hypothesis, two meat products without additives or allergens were produced (cooked ham and cooked turkey breast), and a double-blind, randomised, controlled, unicentric trial with two parallel arms will be conducted.

Prior to the start of the intervention period (baseline time) anthropometric measurements and blood, faeces and urine samples will be taken. 58 participants will take alternately 100g of cooked ham or cooked turkey breast (control or reformulated depending on the group) 6 days a week for 5 weeks, noting the rest of their diet in a collection notebook that they will then give to the researchers. After the intervention (final time), anthropometric measurements and blood, faeces and urine samples will be taken again.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes (men or women) between 18 and 65 years of age
* Body mass index between 18.5 and 30 Kg / m^2.

Exclusion Criteria:

* Diabetes mellitus, chronic kidney disease, liver disease, infectious diseases or any type of cancer.
* Eating disorders, intestinal or similar problems.
* Subjects in treatment with medication for hypertension or hyperlipaemia.
* Subjects in treatment with antibiotics in the last 3 months.
* Subjects who have ingested pre- or probiotic supplements.
* Subjects who have ingested omega-3 or omega-6 supplements.
* Patients undergoing major surgery in the last 3 months prior to the beginning of the study.
* Subjects who have donated blood in the last month prior to the beginning of the study.
* Subjects with alcohol abuse, or with excessive alcohol consumption.
* Vegetarian subjects.
* Pregnant women.
* Smokers.
* Participation in other clinical trials in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Changes in seric lipid profile | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Seric measurement of triglycerides, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C) and total cholesterol.
Changes in serum levels of oxidative stress | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Seric measurement of malondialdehyde (MDA), serum glutathione peroxidase (GPx), catalase (CAT), oxidized LDL, Ferric reducing ability of plasma (FRAP) and ABTS (2,2'-azino-bis(3-methylbenzothiazole-6-sulfonic acid).
Changes in serum levels of inflammation markers | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Seric measurement of C-reactive protein (CRP), Tumor necrosis factor α (TNF-α), Interleukin 1β (IL-1β), Interleukin 6 (IL-6) and Interleukin 10 (IL-10).
Changes in microbiota composition | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Measurement of changes in the abundance of the different bacteria present in the gut.

SECONDARY OUTCOMES:
Serum levels of glucose | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
Serum levels of Alanine Transaminase (ALT) and Aspartate Aminotransferase (AST) | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
Changes in the concentration of nitrates in urine | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
Changes in faecal levels of oxidative stress | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Measurement of FRAP levels in faeces.
Changes in urine levels of oxidative stress | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Measurement of FRAP levels in urine.
Changes in the concentration of short chain fatty acids in faeces. | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
  Measurement of acetate, propionate, butyrate and total SCFA in faeces.
Changes in body mass Index (BMI) | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
Changes in hip-to-waist ratio | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)
Changes in body fat mass percentage | At the beginning of the intervention (baseline) and after 5 weeks of product intake (final time)

CONTACTS AND LOCATIONS:
Locations (1):
- Edificio Pleyades-Vitalys, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT06392893/Prot_ICF_000.pdf